CLINICAL TRIAL: NCT00480428
Title: Study to Improve Thyroid Doses From Fallout Exposure in Kazakhstan
Brief Title: Radiation Exposure and Thyroid Disease in Kazakhstan
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907151; 07-C-N151
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2017-08-17

CONDITIONS: Thyroid Cancer; Thyroid Nodules; Other Thyroid Disease
Keywords: Radioactive Fallout; Childhood Exposures; External Radiation Dose; Internal Radiation Dose to Thyroid Gland; Pasture-Dairy Animal- Milk- Thyroid Pathway
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Residents of certain villages in Kazakhstan were exposed during childhood to radioactive fallout from nuclear tests conducted at the Semipalatinsk Nuclear Test Site (SNTS) between 1949 and 1962.

Radiation doses to the thyroid from external and internal (i.e., ingested) radiation sources deposited as fallout are of interest because they may be jointly and differentially associated with increased risk of thyroid disease in this population.

Objectives:

To collect information about factors influencing radiation dose to the thyroid gland in children of two ethnic groups who were exposed to radioactive fallout from nuclear tests at the SNTS between 1949 and 1962. The two groups are Kazakhs (historically nomadic herders) and Europeans (typically descendants of Russian and German farmers).

Eligibility:

Women 70 years of age and older who had children or provided care to children during the 1950s.

Men age 70 and older who were engaged in farming and care of dairy animals at the time of the nuclear tests.

Design:

In focus group format, participants are interviewed to collect information on the following at the time of nuclear tests:

* Dairy consumption;
* Source, storage and availability of milk and milk products;
* Time that children of different ages and ethnic groups spent indoors;
* Building material of houses and schools;
* Herding, grazing and supplemental feed of dairy animals.

DETAILED DESCRIPTION:
The proposed work will improve our understanding of historical, fallout-related radiation doses received by residents of villages in Kazakhstan immediately downwind from the Semipalatinsk Nuclear Test Site (SNTS), where multiple nuclear test explosions were carried out between 1949 and 1962. In collaboration with scientists at the Institute for Biophysics in Moscow, NCI has developed a combined bi-national dose reconstruction methodology based on lessons learned from studying radioactive fallout from tests at the SNTS in Kazakhstan, the Nevada Test Site in the United States, and other test sites. Gamma rays from radionuclides such as cesium 137 in fallout are highly penetrating and can affect all organs even when the radioactive source is outside the body, whereas less-penetrating beta particles from iodine 131, also plentiful in fallout, mainly affect the thyroid gland when ingested in milk from dairy animals grazing on contaminated pasture. We are particularly interested in both kinds of radiation doses to children, because their thyroid glands are small and very active, tend to concentrate ingested iodine, and are highly sensitive to radiation carcinogenesis. The conditions of fallout exposure in Kazakhstan are directly relevant to those following a hypothetical nuclear accident or radiation terrorism incident involving high levels of local fallout.

We propose a field study in Kazakhstan to investigate aspects of typical daily village life in areas affected by fallout that might influence individual radiation doses to the thyroid gland. Using focus group interviews, we will collect retrospective information about factors influencing radiation dose to the thyroid gland in children of two distinct ethnic groups (Kazakh and European). These factors include milk and milk product consumption, dependence on different species of dairy animals known to differ with respect to concentration of iodine in milk, seasonal practices of pasturing and supplemental feeding of dairy animals at the time of the nuclear tests, time children typically spent outdoors, and radiation shielding provided by dwellings and other buildings. We will also ask about protective measures taken at the time, such as details of temporary evacuations of villages predicted to be in the fallout paths from particular tests. These data will fill key gaps in the current dose-reconstruction methodology and should result in improved dose estimates, as well as a basis for evaluating and quantifying dosimetric uncertainty and related biases in risk estimates.

ELIGIBILITY:
* To be eligible, individuals must speak Russian or Kazakh, be able to participate in a two-hour focus group session, and have a verified history of residing in the village during the 1950s. Verification of residence history will be based on regional records.

  1. Women: In each village, we will recruit 24 women. We will select women who are age 70 years and older and who had children or provided care to children (i.e., younger siblings, nieces and nephews) during the 1950s. Our first priority is to recruit women whose own children were less than 21 years during the 1950s. If necessary, we will also recruit women who provided care to children other than their own (e.g., younger siblings, nieces and nephews) during this period. We will recruit both members of our 1998 cohort members and other women in the community who meet the eligibility criteria. Subjects will be chosen to represent experience caring for children of different ages at the time of the nuclear tests. In order to recruit women who had children of different ages (less than 21 years) during the 1950s, we will screen potential participants for their children s years of birth and attempt to enroll women whose children represent a range of ages during the 1950 s.
  2. Men: In each village, we will recruit eight men (Russian and Kazakh) age 70 and older who were engaged in farming and care of dairy animals at the time of the nuclear tests.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 117 (Actual)
Dates: Start 2007-05-17; Study Completion 2017-08-17

PRIMARY OUTCOMES:
Thyroid nodules | 1998

CONTACTS AND LOCATIONS:
Overall Officials: Kiyohiko Mabuchi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Semipalatinsk State Medical Academy, Semipalatinsk, Kazakhstan

REFERENCES:
- [Background] Anspaugh LR, Simon SL, Gordeev KI, Likhtarev IA, Maxwell RM, Shinkarev SM. Movement of radionuclides in terrestrial ecosystems by physical processes. Health Phys. 2002 May;82(5):669-79. doi: 10.1097/00004032-200205000-00013. PMID 12003017
- [Background] Degteva MO, Vorobiova MI, Tolstykh EI, Shagina NB, Shishkina EA, Anspaugh LR, Napier BA, Bougrov NG, Shved VA, Tokareva EE. Development of an improved dose reconstruction system for the Techa River population affected by the operation of the Mayak Production Association. Radiat Res. 2006 Jul;166(1 Pt 2):255-70. doi: 10.1667/RR3438.1. PMID 16808612
- [Background] Bogdanova TI, Zurnadzhy LY, Greenebaum E, McConnell RJ, Robbins J, Epstein OV, Olijnyk VA, Hatch M, Zablotska LB, Tronko MD. A cohort study of thyroid cancer and other thyroid diseases after the Chornobyl accident: pathology analysis of thyroid cancer cases in Ukraine detected during the first screening (1998-2000). Cancer. 2006 Dec 1;107(11):2559-66. doi: 10.1002/cncr.22321. PMID 17083123